CLINICAL TRIAL: NCT06497855
Title: Impact of Target Controlled Infusion Estimated Concentration of Propofol on Implicit Memory Formation During Propofol-Remifentanil General Anaesthesia
Brief Title: Impact of Estimated Concentration of Propofol on Implicit Memory Formation
Status: Not yet recruiting | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Other Study IDs: ImpliMAST
Record Dates: First submitted 2024-07-01; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-06

CONDITIONS: General Anaesthesia; Implicit Memory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients who, during general anaesthesia, will hear the 20 words and will be tested form implicit memory formation.
- Controls: Patients who, during general anaesthesia, will not hear the 20 words and will be tested form implicit memory formation to assess the role of chance on the tests adopted

SUMMARY:
Implicit memory formation and learning during general anaesthesia is a still debated question and no anesthetic regimen (ie intravenous anaesthesia vs inhalatory one) nor analgesic regimen (i.e. low or high opioids usage) has been identified for prevention.

With this study the investigators aim to investigate if, during Total Intravenous Anaesthesia with Target Controlled Infusion (TIVA-TCI) different concentrations of Propofol at loss of responsiveness, maintenance and return of responsiveness can have a role in implicit memory formation.

DETAILED DESCRIPTION:
Implicit memory formation and learning during general anaesthesia is a still debated question and no anesthetic regimen (ie intravenous anaesthesia vs inhalatory one) nor analgesic regimen (i.e. low or high opioids usage) has been identified for prevention.

With this study the investigators aim to investigate if, during Total Intravenous Anaesthesia with Target Controlled Infusion (TIVA-TCI) different concentrations of Propofol at loss of responsiveness (CeP RoR), maintenance (CePMA) and return of responSiveness (CeP RoR) can have a role in implicit memory formation.

20 most common italiaN words will be continuously presented to the anaesthetized patients from Loss of responsiveness to end of surgery.

CeP RoR, MA and LoR, as well as patient state index (PSi) from Sedline monitor for hypnosis level monitoring will be recorded.

Within 24 hours, a trained psychologist will be present the patients the Word Steam Recognition Test, Free Recall and Force Choice recognition task to asses the presence of implicit memory formation. A second group, who did not hear the words, will be investigated to assess the role of chance in the above-mentioned test.

ELIGIBILITY:
Inclusion Criteria:

* General anaesthesia with TIVA-TCI

Exclusion Criteria:

* ASA > III
* Benzodiazepines premedication
* Neurological/Psychiatric disease

Ages: 18 Years to 90 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Breast-Surgery women undergoing TIVA-TCI
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
The role of Propofol Concentration at the loss of responsiveness on Implicit Memory formation | CeP will be recorded at Loss of responsiveness. Word Steam recognition, Free recall and Forced Choice Recognition Task will be performed within 12-24 hours after surgery. These 3 tests are analysed togheter to check for implicit memory formation.
  CeP at LOR will be compared between patients who exhibit or not implicit memory formation.
The role of Propofol Concentration at the maintenance of anaesthesia on Implicit Memory formation | CeP will be recorded during anaesthesia maintenance. Word Steam recognition, Free recall and Forced Choice Recognition Task will be performed within 12-24 hours after surgery. These 3 tests are analysed togheter to check for implicit memory formation.
  CeP at anaesthesia maintenance will be compared between patients who exhibit or not implicit memory formation.
The role of Propofol Concentration at the return of responsiveness on Implicit Memory formation | CeP will be recorded at Return of responsiveness. Word Steam recognition, Free recall and Forced Choice Recognition Task will be performed within 12-24 hours after surgery. These 3 tests are analysed togheter to check for implicit memory formation.
  CeP at ROR will be compared between patients who exhibit or not implicit memory formation.